CLINICAL TRIAL: NCT02339285
Title: Pilot Clinical Trial for the Evaluation of Feedback Transcranial Alternating Current Stimulation for the Treatment of Major Depressive Disorder
Brief Title: Transcranial Alternating Current Stimulation for Major Depressive Disorder
Acronym: MDD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 14-1622; 5R01MH101547-02 (NIH)
Record Dates: First submitted 2015-01-12; First posted 2015-01-15 (Estimated); Results first posted 2018-08-20 (Actual); Last update posted 2018-08-20 (Actual); Status verified 2018-01

CONDITIONS: Major Depressive Disorder; MDD
Keywords: tACS; Major Depressive Disorder; MDD; mood symptoms; sham
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- tACS (alpha) (Experimental): 10 Hz tACS with a peak-to-peak amplitude of 2 milliamps (mA) for 40 minutes. Uses tACS (alpha) device.
  Interventions: Device: tACS (alpha)
- tACS (gamma) (Experimental): 40 Hz tACS with a peak-to-peak amplitude of 2 milliamps (mA) for 40 minutes. Uses tACS (gamma) device.
  Interventions: Device: tACS (gamma)
- Sham stimulation (Sham Comparator): Will include 10 seconds of ramp in to 1 minute of 10 Hz tACS with a ramp out of 10 seconds for a total of 80 seconds of stimulation. Uses tACS (alpha) device.
  Interventions: Device: tACS (alpha)

INTERVENTIONS:
Device: tACS (alpha)
  Arms: Sham stimulation; tACS (alpha)
Device: tACS (gamma)
  Arms: tACS (gamma)

SUMMARY:
Investigating the effects of non-invasive transcranial alternating current stimulation (tACS) on patients with Major Depressive Disorder (MDD).

DETAILED DESCRIPTION:
Central Hypothesis: Non-invasive brain stimulation that suppresses alpha oscillation reduces cortical hyperactivity and causes a clinical improvement

Aim 1: To conduct a pilot clinical trial to establish feasibility and to collect first effectiveness data for the use of tACS to renormalize pathological alpha oscillations in the dorsolateral prefrontal cortex (dl-pfc) of unmedicated patients with MDD by comparing MADRS scores from baseline and one month follow up.

Aim 2: Compare alpha oscillation power from resting state EEG recordings on the first and last day of stimulation. Collect EEG data at the one month follow up visit using this data to analyze alpha frequency activity as a pilot study for derivation of EEG biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, 18-65 years old
* Diagnostic and Statistical Manual of Mental Disorder, 4th edition (DSM-IV) diagnosis of MDD; unipolar, non-psychotic
* Hamilton Depression Rating Scale score >8
* Capacity to understand all relevant risks and potential benefits of the study (informed consent)
* Meet criteria for low suicide risk
* Willing to comply with all study procedures and be available to do so for the duration of the study
* Women of reproductive potential must use highly effective contraception

Exclusion Criteria:

* DSM-IV diagnosis of alcohol of substance abuse (other than nicotine) within the last month or a DSM-IV diagnosis of alcohol or substance dependence (other than nicotine) within the last 6 months
* Current use of benzodiazepines or anti-epileptic drugs
* Current axis I mood, or psychotic disorder other than major depressive disorder
* Lifetime comorbid psychiatric bipolar or psychotic disorder
* Eating disorder (current or within the past 6 months)
* Obsessive-compulsive disorder (lifetime)
* Post traumatic stress disorder (PTSD; current or within the last 6 months)
* Attention Deficit Hyperactivity Disorder (ADHD; currently under treatment)
* Anything that, in the opinion of the investigator, would place the participant at increased risk or preclude the participant's full compliance with or completion of the study
* Neurological disorders, including but not limited to history of seizures (except childhood febrile seizures and ECT induced seizures), dementia, history of stroke, Parkinson's disease, multiple sclerosis, cerebral aneurism
* Medical or neurological illness (unstable cardiac disease, AIDS, malignancy, liver or renal impairment) or treatment for a medical disorder that could interfere with study participation
* History of traumatic brain injury, reoccurring seizures or later cognitive rehabilitation, or causing cognitive sequelae
* Prior brain surgery
* Any brain devices/implants, including cochlear implants and aneurysm clips
* Co-morbid neurological condition (i.e. seizure disorder, brain tumor)
* Non English speakers
* Pregnancy, nursing, or if female and fertile, unwilling to use appropriate birth control measures during study participation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2015-05-07 (Actual); Primary Completion 2017-06-19 (Actual); Study Completion 2017-06-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Flavio Frohlich, PhD, Principal Investigator — University of North Carolina at Chapel Hill, Department of Psychiatry
Locations (1):
- UNC Chapel Hill Medical School Wing C, Chapel Hill, North Carolina, United States

REFERENCES:
- [Background] Valiengo L, Bensenor IM, Goulart AC, de Oliveira JF, Zanao TA, Boggio PS, Lotufo PA, Fregni F, Brunoni AR. The sertraline versus electrical current therapy for treating depression clinical study (select-TDCS): results of the crossover and follow-up phases. Depress Anxiety. 2013 Jul;30(7):646-53. doi: 10.1002/da.22079. Epub 2013 Apr 26. PMID 23625554

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited through advertisements (e.g., online, flyers) and self-identified with depression. Interested participants contacted the study team.
Pre-assignment Details: Participants were randomly assigned to 1 of 3 arms: tACS (alpha), tACS (gamma), or sham stimulation. All conditions were delivered during awake, resting state for 40 minutes on 5 consecutive days. 98 participants signed consent, 40 did not meet criteria, 6 declined participation, and 20 were excluded for other reasons. 32 were randomized.
Groups:
- tACS (Alpha): 10 Hz transcranial alternating current stimulation (tACS) with a peak-to-peak amplitude of 2 mA for 40 minutes
- tACS (Gamma): 40 Hz transcranial alternating current stimulation with a peak-to-peak amplitude of 2 mA for 40 minutes
- Sham Stimulation: Will include 10 seconds of ramp in to 1 minute of 10 Hz tACS with a ramp out of 10 seconds for a total of 80 seconds of stimulation.
Period: Overall Study
Arm/Group | tACS (Alpha) | tACS (Gamma) | Sham Stimulation
Started (All randomized participants included in analysis. Intent-to-treat; last observation carried forward.) | 10 | 11 | 11
Completed Intervention (Number of participants that completed 5 days of stimulation.) | 10 | 10 | 10
2 Week Follow-up (Number of participants that attended the follow-up visit 2 weeks after completion of intervention.) | 9 | 10 | 10
4 Week Follow-up Visit (Number of participants that attended the follow-up visit 4 weeks after completion of intervention.) | 9 | 8 | 9
Completed (Number of participants that completed all sessions.) | 9 | 8 | 9
Not Completed | 1 | 3 | 2
Not completed — Withdrawal by Subject | 0 | 1 | 1
Not completed — Lost to Follow-up | 1 | 1 | 1
Not completed — Protocol Deviation | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- tACS (Alpha): 10 Hz transcranial alternating current stimulation with a peak-to-peak amplitude of 2 mA for 40 minutes
- Total: Total of all reporting groups
Arm/Group | tACS (Alpha) | tACS (Gamma) | Sham Stimulation | Total
Number analyzed (Participants) | 10 | 11 | 11 | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.30 (15.22) | 35.36 (11.56) | 38.36 (13.54) | 36.69 (13.08)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 9 | 9 | 27
  Male | 1 | 2 | 2 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 6 | 10 | 10 | 26
  Unknown or Not Reported | 4 | 1 | 1 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 1
  Asian | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 9 | 10 | 11 | 30
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 10 | 11 | 11 | 32
Montgomery-Asberg Depression Rating Scale (MADRS) [Mean (Standard Deviation); unit: units on a scale] — The MADRS is a 10-item scale to measure the severity of depressive episodes, where each item is rated on a scale from 0 to 6. The MADRS total score ranges from 0 to 60 with lower scores indicating less depressive symptoms.
  units on a scale | 28.80 (6.36) | 25.00 (7.21) | 24.55 (5.18) | 26.03 (6.39)
Hamilton Depression Rating Scale (HDRS) [Mean (Standard Deviation); unit: units on a scale] — The HDRS is a clinician-administered depression assessment and consists of 17 items with a total score range from 0 to 54. Higher scores indicate more depressive symptoms.
  units on a scale | 17.90 (4.51) | 14.64 (3.53) | 14.55 (6.12) | 15.63 (4.94)
Beck Depression Inventory (BDI) [Mean (Standard Deviation); unit: units on a scale] — The BDI is a self-administered questionnaire that measures the occurrence and severity of current depressive symptoms. Total scores range from 0-63 with higher scores indicating higher feelings of being depressed.
  units on a scale | 26.60 (5.58) | 28.27 (8.81) | 26.18 (9.74) | 27.03 (8.10)
Montreal Cognitive Assessment (MoCA) [Mean (Standard Deviation); unit: units on a scale] — A basic assessment of cognition. Total score is ranges from 0 to 30 points, with higher values indicating better cognition.
  units on a scale | 28.20 (1.99) | 27.27 (1.62) | 27.82 (2.48) | 27.75 (2.00)
Clinical Global Impression (CGI) [Mean (Standard Deviation); unit: units on a scale] — Values reported on Item 1 "Severity of Illness" on the Clinical Global Impressions scale. Patients are scored on a likert scale, with 1 = "Normal, not at all ill" to 7 = "Among the most extremely ill patients."
  units on a scale | 4.10 (0.99) | 3.82 (0.60) | 3.73 (0.79) | 3.88 (0.79)

OUTCOME MEASURES:

1. Primary Outcome: Change in the Montgomery-Asberg Depression Rating Scale (MADRS) Score
Description: The MADRS is a 10-item scale to measure the severity of depressive episodes, where each item is rated on a scale from 0 to 6. The MADRS total score ranges from 0 to 60 with lower scores indicating less depressive symptoms. This measurement will be taken at baseline (Day 1 of Stimulation), Day 5 of Stimulation, 2 weeks after completion of the intervention (F1), and 4 weeks after completion of the intervention (F2). A comparison of MADRS scores between baseline and F2 is the primary outcome measure (measured as change from baseline). In these results, negative values will indicate a decrease in depressive symptoms.
Time Frame: Baseline to F2 (4 weeks after completion of the intervention)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | tACS (Alpha) | tACS (Gamma) | Sham Stimulation
Number analyzed (Participants) | 10 | 11 | 11
units on a scale | -13.60 (7.75) | -8.82 (8.94) | -8.27 (10.88)
Statistical Analysis 1: Comparison: tACS (Alpha) vs tACS (Gamma) vs Sham Stimulation; Null hypothesis: There is no difference baseline and the 4 week follow up in MADRS score between treatment groups. Alternative hypothesis: There is a difference between baseline and the 4 week follow up MADRS score between treatment groups; Test type: Other — F-test; Treatment effect; p > 0.10, ANOVA; F(2, 29)
Statistical Analysis 2: Comparison: tACS (Alpha) vs tACS (Gamma) vs Sham Stimulation; [analysis description as in outcome 1, analysis 1]; Test type: Other — F-test; Session effect; p < 0.001, ANOVA; F(1, 31)
Statistical Analysis 3: Comparison: tACS (Alpha) vs tACS (Gamma) vs Sham Stimulation; Test type: Other — F-test; Interaction effect (session x treatment); p > 0.10, ANOVA; F(2,29)

2. Secondary Outcome: Change in Alpha Oscillation Power From Resting State EEG Recordings on the First and Last Day of Stimulation
Description: The investigators will compare alpha oscillation power from resting state EEG recordings on the first day of stimulation (baseline) and last day of stimulation. The investigators will also collect EEG recordings data at a visit four weeks after completion of the intervention (F2). The investigators will use each of the three EEG recordings as data to analyze alpha frequency activity as a pilot study for derivation of EEG biomarkers. As the stimulation paradigm stimulates the frontal brain regions, the investigators will analyze alpha power change in all brain regions as well as frontal regions.
Time Frame: Baseline to Day 5 of Stimulation
Population: Only participants that completed all sessions are used in this task (per protocol participants); N = 26
Measure: Mean (Standard Deviation); unit: decibel (dB)
Arm/Group | tACS (Alpha) | tACS (Gamma) | Sham Stimulation
Number analyzed (Participants) | 9 | 8 | 9
decibel (dB)
  All Brain Regions | -1.75 (1.75) | 0.53 (1.79) | 0.24 (1.22)
  Frontal Brain Regions | -1.23 (1.29) | 0.12 (1.68) | -0.02 (1.20)
Statistical Analysis 1: Comparison: tACS (Alpha) vs tACS (Gamma) vs Sham Stimulation; Null hypothesis: There is no difference in changes of alpha frequency power between baseline EEG and EEG on Day 5 of Stimulation between treatment groups. Alternative hypothesis: There is a difference in changes of alpha frequency power between baseline EEG and EEG on Day 5 of Stimulation between treatment groups; Test type: Other — F-test; Condition effect; p < 0.05, ANOVA; F(2,21.595)
Statistical Analysis 2: Comparison: tACS (Alpha) vs tACS (Gamma) vs Sham Stimulation; [analysis description as in outcome 2, analysis 1]; Test type: Other — F-test; Region effect (region defined as region of brain - frontal, parietal, occipital temporal); p < 0.001, ANOVA; F(3, 79.358)
Statistical Analysis 3: Comparison: tACS (Alpha) vs tACS (Gamma) vs Sham Stimulation; [analysis description as in outcome 2, analysis 1]; Test type: Other — F-test; Interaction effect (region x condition); p > 0.10, ANOVA; F(6, 68.284)

3. Secondary Outcome: Change in Alpha Oscillation Power From Resting State EEG Recordings on the First of Stimulation to 4 Weeks After Completion of Intervention
Description: The investigators will compare alpha oscillation power from resting state EEG recordings on the first day of stimulation (baseline) and at the follow-up visit four weeks after completion of the intervention. The investigators will also collect EEG on the fifth day of stimulation. The investigators will use each of the three EEG recordings as data to analyze alpha frequency activity as a pilot study for derivation of EEG biomarkers. As the stimulation paradigm stimulates the frontal brain regions, the investigators will analyze alpha power change in all brain regions as well as frontal regions.
Time Frame: Baseline to F2
Population: Only participants that completed all sessions are used in this task (per protocol participants); N = 26
Measure: Mean (Standard Deviation); unit: decibel (dB)
Arm/Group | tACS (Alpha) | tACS (Gamma) | Sham Stimulation
Number analyzed (Participants) | 9 | 8 | 9
decibel (dB)
  All Brain Regions | -0.42 (2.35) | 0.09 (1.76) | 0.55 (1.17)
  Frontal Brain Regions | -0.57 (1.89) | 0.00 (1.60) | 0.41 (1.18)
Statistical Analysis 1: Comparison: tACS (Alpha) vs tACS (Gamma) vs Sham Stimulation; Null hypothesis: There is no difference in changes of alpha frequency power between baseline EEG and EEG 4 weeks after completion of the intervention between treatment groups. Alternative hypothesis: There is a difference in changes of alpha frequency power between baseline EEG and EEG 4 weeks after completion of the intervention between treatment groups; Test type: Other; p > 0.10, ANOVA

4. Other Pre Specified Outcome: Change in Hamilton Depression Rating Scale (HDRS) Score
Description: The HDRS is a clinician-administered depression assessment and consists of 17 items with a total score range from 0 to 54. A higher score indicates a worse outcome. This measurement will be taken at baseline (Day 1 of Stimulation), Day 5 of Stimulation, 2 weeks after completion of the intervention (F1), and 4 weeks after completion of the intervention (F2). The investigators will compare the scores between baseline and F2, with negative values indicating a decrease in depressive symptoms.
Time Frame: Baseline to Day 5 of Stimulation; Baseline to F2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | tACS (Alpha) | tACS (Gamma) | Sham Stimulation
Number analyzed (Participants) | 10 | 11 | 11
units on a scale
  Day 5 change | -6.00 (3.09) | -4.45 (5.41) | -3.09 (4.48)
  F2 change | -8.50 (5.04) | -4.73 (5.61) | -4.64 (6.98)

5. Other Pre Specified Outcome: Change in Montreal Cognitive Assessment (MoCA) Score
Description: This measurement will be taken at baseline (first day of stimulation) and four weeks after completion of the intervention (F2). Total score ranges from 0 to 30, with higher values indicating better cognition. The investigators will compare the scores between baseline and F2. Reported values are the raw change (increase or decrease) from baseline.
Time Frame: Baseline to F2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | tACS (Alpha) | tACS (Gamma) | Sham Stimulation
Number analyzed (Participants) | 10 | 11 | 11
units on a scale | 0.50 (0.53) | 1.27 (1.35) | 1.09 (1.51)

6. Other Pre Specified Outcome: Change in Beck Depression Inventory (BDI) Score
Description: This measurement will be taken at baseline (Day 1 of Stimulation), Day 5 of Stimulation, 2 weeks after completion of the intervention (F1), and 4 weeks after completion of the intervention (F2). Higher scores indicate more depressive symptoms. Total score is out of 63 possible. The investigators will compare the scores between baseline and F2. In these results, negative values indicate a decrease in depressive symptoms.
Time Frame: Baseline to Day 5; Baseline to F2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | tACS (Alpha) | tACS (Gamma) | Sham Stimulation
Number analyzed (Participants) | 10 | 11 | 11
units on a scale
  Day 5 Change | -8.60 (6.42) | -9.64 (10.07) | -7.18 (7.19)
  F2 change | -14.80 (12.39) | -11.09 (11.68) | -10.64 (10.39)

7. Other Pre Specified Outcome: Clinical Global Impressions (CGI) Raw Score
Description: This measurement will be taken at baseline (Day 1 of Stimulation), Day 5 of Stimulation, 2 weeks after completion of the intervention (F1), and 4 weeks after completion of the intervention (F2). The investigators will compare the scores between baseline and F2.The reported values are from Item 1 "Severity of Illness" on a likert scale of 1 to 7, with 1=Normal, not at all ill and 7 = Among the most extremely ill patients.
Time Frame: Day 5; F2 (4 weeks after completion of treatment)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | tACS (Alpha) | tACS (Gamma) | Sham Stimulation
Number analyzed (Participants) | 10 | 11 | 11
units on a scale
  Day 5 Score | 4.30 (0.95) | 3.73 (0.65) | 3.73 (0.79)
  F2 Score | 3.90 (1.37) | 3.82 (0.75) | 3.45 (1.29)

ADVERSE EVENTS:
Time Frame: Throughout the intervention period and throughout F2 (4 weeks after completion of the intervention), for an average of 5 weeks.
Arm/Group | tACS (Alpha) | tACS (Gamma) | Sham Stimulation
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/11 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/11 | 0/11
Other Adverse Events (participants affected / at risk) | 0/10 | 0/11 | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-01-04): https://cdn.clinicaltrials.gov/large-docs/85/NCT02339285/Prot_SAP_000.pdf